CLINICAL TRIAL: NCT00881218
Title: Feasibility of Detecting Myocardial Ischemia by First-pass Contrast MRI Using Regadenoson
Brief Title: Myocardial Perfusion Magnetic Resonance Imaging Using Regadenoson
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Pamela Woodard, MD, M.D., FACR, FAHA, FCCP, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: REGADENOSON.MRI.WUSTL
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Ischemic Heart Disease
Keywords: myocardial ischemia, perfusion imaging, cardiac MRI
MeSH Terms: conditions — Myocardial Ischemia | interventions — regadenoson

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regadenoson CMR (Experimental): Images in the cardiac short axis will be obtained using a gradient recalled echo sequence, TR 2.3 msec/TE 1.1 msec, 80*256 matrix, slice thickness 10 mm. Images will be obtained during power injection of 0.075 mmol/Kg of a conventional gadolinium based MR contrast agent at a rate of 5 mL/sec followed by a 15 mL saline flush into an antecubital vein. Perfusion imaging will be performed at stress and rest. Stress: Regadenoson 400 mcg will be administered IV bolus via an antecubital cannula. Immediately after injection, MR scanning will begin and contrast will be given. Rest: After 10 minutes, rest imaging will be performed identically, but without regadenoson injection. To identify late enhancement of myocardial tissue inversion recovery prepared images will be obtained.
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — Regadenoson 400 micrograms will be administered IV bolus via an antecubital cannula.
  Other Names: Lexiscan

SUMMARY:
This is a pilot study to determine whether the drug regadenoson can be used during magnetic resonance imaging to assess regions of poor blood flow to the heart.

The hypothesis of this study is that a single injection of regadenoson could be used instead of a standard adenosine infusion to produce coronary vasodilatation and demonstrate myocardial ischemia during first-pass perfusion cardiac MRI.

DETAILED DESCRIPTION:
This is a pilot study that proposes to assess the feasibility of using regadenoson (Lexiscan, Astellas), a recently FDA approved A2A receptor agonist, as the stress perfusion agent in cardiac MRI perfusion examinations. While regadenoson has been approved by the FDA, it has not been approved for the specific indications of use 1) during the simultaneous intravenous administration of a gadolinium-based contrast agent, or 2) during magnetic resonance imaging (MRI).

Because this agent can be given intravenously in a single 400 microgram bolus, rather than in an infusion, this agent may be easier to administer than adenosine during an MRI examination.

The objectives for this pilot study are: 1) To demonstrate the feasibility of using regadenoson during cardiac perfusion MRI to visualize known regions of myocardial ischemia as demonstrated on SPECT-MPI and 2) To describe a cardiac perfusion MRI protocol using regadenoson that would have the potential to be used clinically.

ELIGIBILITY:
Inclusion Criteria:

* reversible perfusion abnormalities on a clinically ordered rest/adenosine dual-isotope SPECT-MPI in at least 2 contiguous myocardial segments (per 17-segment model)

Exclusion Criteria:

* myocardial infarction, myocardial revascularization procedure or progression in angina occuring after the SPECT-MPI examination
* pregnancy
* gadolinium-based MR contrast allergy
* glomerular filtration rate (GFR) > 60 mL/min/1.73 m2
* contraindications to MR imaging (pacemaker, brain aneurysm clips, schrapnel, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of use of regadenoson during cardiac perfusion MRI to visualize regions of myocardial ischemia as demonstrated on SPECT-MPI. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K. Woodard, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Aljaroudi W, Hermann D, Hage F, Heo J, Iskandrian AE. Safety of regadenoson in patients with end-stage renal disease. Am J Cardiol. 2010 Jan 1;105(1):133-5. doi: 10.1016/j.amjcard.2009.08.663. Epub 2009 Nov 18. PMID 20102905
- [Background] Iskandrian AE, Bateman TM, Belardinelli L, Blackburn B, Cerqueira MD, Hendel RC, Lieu H, Mahmarian JJ, Olmsted A, Underwood SR, Vitola J, Wang W; ADVANCE MPI Investigators. Adenosine versus regadenoson comparative evaluation in myocardial perfusion imaging: results of the ADVANCE phase 3 multicenter international trial. J Nucl Cardiol. 2007 Sep-Oct;14(5):645-58. doi: 10.1016/j.nuclcard.2007.06.114. PMID 17826318
- [Background] Cerqueira MD, Nguyen P, Staehr P, Underwood SR, Iskandrian AE; ADVANCE-MPI Trial Investigators. Effects of age, gender, obesity, and diabetes on the efficacy and safety of the selective A2A agonist regadenoson versus adenosine in myocardial perfusion imaging integrated ADVANCE-MPI trial results. JACC Cardiovasc Imaging. 2008 May;1(3):307-16. doi: 10.1016/j.jcmg.2008.02.003. PMID 19356442